CLINICAL TRIAL: NCT05900128
Title: Impact of Exercise on Asthma Control and Management in Adults
Brief Title: Impact of Exercise on Ashtma in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EC075-23_HRJC
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-04

CONDITIONS: Asthma; Physical Inactivity
Keywords: asthma; sedentarism; spirometry; physical excercise
MeSH Terms: conditions — Asthma; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): asthmatic patients who receive the educative intervention
  Interventions: Behavioral: workshop
- no intervention (Placebo Comparator): asthmatic patients who don't receive the educative intervention
  Interventions: Other: no workshop

INTERVENTIONS:
Behavioral: workshop — Patients will receive workshops and they will encourage to practice physical activity
  Arms: Intervention
Other: no workshop — patients won't receive educative workshops
  Arms: no intervention

SUMMARY:
The aim of this study is to evaluate if physical activity could improve asthma control and management in adults. With this purpose we enroll asthmatic patients between 18-64 years old, and randomized them into 2 groups: in the first, patients will receive some workshops about asthma en physical exercise; in the second no educational intervention will be done. All patients will use a step counter in order to evaluate their activity during the study. Spirometric values and questionnaries about asthma control and quality of life will be recorded for all patients. Finally 2 groups will be comparated in order to search any difference in quality of life and asthma control.

DETAILED DESCRIPTION:
52 asthmatic will be enrolled and randomized into 2 groups. All patients will send a weekly summary of their physical activity (mean number of steps and time of physical activity). All patients will be undergone to a medical visit at month 1 and 3 since study start. In each visit a spirometry, a FeNo, ACQ and AQLQ questionnaires will be done.

The patients of the intervention group will receive 3 workshops about asthma and physical exercise in order to provide information, medical support, and to resolve any question or difficulty about it. The workshops will be al week 1, 2 and 4 since study start.

ELIGIBILITY:
Inclusion Criteria:

* asthma well controlled
* sedentarism (<150 min physical activity/day and/or <7000 daily steps)

Exclusion Criteria:

* pregnancy
* cardiological, not well controlled deseases
* other cronic pulmonary deseases
* bad asthma control
* not sign IC
* unable to practice physical activity (for cognitive or physical conditions)
* no devices able to count steps and physical activity

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Improvement of asthma control | 3 months
  change of 0.5 points in Asthma Control Questionnaire (0-6; higher score means worse result)

CONTACTS AND LOCATIONS:
Overall Officials: sarah micozzi, MD, Principal Investigator — Hospital Rey Juan Carlos-Instituto de Investigación FJD
Locations (1):
- Hospital Rey Juan Carlos, Móstoles, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Pending to decide if share the final report with other researchers